CLINICAL TRIAL: NCT02068365
Title: An Open-label Trial of 48-week Peginterferon Alfa-2a (PEGASYS) to Assess the Sustained Response of Chronic Hepatitis B Patients With HBeAg Seroconversion on Nucleot(s)Ide Analogue Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Henry LY Chan, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28486
Record Dates: First submitted 2014-01-28; First posted 2014-02-21 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Chronic Hepaititis B

ARMS (1):
- Pegyinterferon-alfa-2a (Other): Pegyinterferon-alfa-2a 180mcq weekly for 48 weeks
  Interventions: Drug: Pegyinterferon-alfa-2a

INTERVENTIONS:
Drug: Pegyinterferon-alfa-2a — Pegyinterferon-alfa-2a 180mcq weekly for 48 weeks

SUMMARY:
This is a multi-center, single-arm, open-label study on the virological response of chronic HBV infection to pegyinterferon-alfa-2a among patients who achieved HBeAg seroconversion on nucleos(t)ide analogue (NA) treatment. The primary endpoint of this study is to investigate the sustained response (HBeAg seroconversion with HBV DNA <2000 IU/ml) to peginterferon at 24 weeks after the end of treatment.

DETAILED DESCRIPTION:
Chronic hepatitis B is the commonest cause of liver cirrhosis and hepatocellular carcinoma in Hong Kong. Treatment with interferon and nucleos(t)ide analogues (NA) can reduce the risk of HCC. NA is the commonest used medication in Hong Kong. However, most patients require long-term treatment and premature drug cessation may lead to hepatitis relapse.

Under the current regional guidelines, patients who have positive hepatitis B e antigen (HBeAg) treated by NA can consider stopping treatment if HBeAg seroconversion has developed for at least 12 months. However, up to 30-50% of patients may develop virological relapse and/or HBeAg reversion after cessation of treatment. On the other hand, interferon-based treatment has a much more durable response. HBeAg seroconversion is maintained in 80% of patients after successful treatment with peginterferon. Upon long-term follow-up, peginterferon-treated patients are also more likely to achieve hepatitis B surface antigen (HBsAg) seroclearance, a condition closest to a cure of chronic hepatitis B.

ELIGIBILITY:
Inclusion Criteria:

* Male & female patients >= 18 and < 70 years of age
* Positive HBeAg before starting NA treatment
* Treated by a single NA (lamivudine, adefovir, entecavir or tenofovir) for 6 months to 5 years
* Developed HBeAg seroconversion (HBeAg negative and ant-HBe negative) with undetectable HBV DNA by PCR based assay on NA treatment.
* Negative urine or serum pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of test drug. Additionally, all females must be using reliable contraception during the study and for 3 months after treatment completion

Exclusion Criteria:

* Evidence of decompensated liver disease (Childs B-C), hepato-cellular carcinoma, pre-existing severe depression or other psychiatric disease, significant cardiac disease, significant renal disease, seizure disorders or severe retinopathy.
* received telbivudine as the antiviral therapy or have received more than one NA in the past.
* received interferon or peginterferon treatment in the past.
* received antiviral therapy for any systemic anti-viral, anti-neoplastic or immuno-modulatory treatment (including supraphysiologic doses of steroids and radiation) within the past 6 months.
* Positive test at screening for anti-HIV, anti-HCV.
* Patients who are expected to need systemic antiviral therapy other than that provided by the study at any time during their participation in the study are also excluded. Exception: patients who have had a limited (<=7 days) course of acyclovir for herpetic lesions more than 1 month prior to the first administration of test drug are not excluded.
* Serum total bilirubin > 3 times the upper limit of normal at screening.
* History or other evidence of bleeding from esophageal varices or other conditions consistent with decompensated liver disease.
* History or other evidence of a medical condition associated with chronic liver disease other than HBV (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver diseases including Wilson's and alpha1-antitrypsin deficiency, alcoholic liver disease, toxin exposures, thalassemia).
* Women with ongoing pregnancy or who are breast feeding.
* Neutrophil count <1500 cells/mm3 or platelet count <90,000 cells/mm3 at screening.
* Hemoglobin < 11.5 g/dL for females and < 12.5 g/dL for men at screening.
* Serum creatinine level >120 umol/ml for men and >105 umol/ml for women at screening.
* History of severe psychiatric disease, especially depression. Severe psychiatric disease is defined as major depression or psychosis, a period of treatment with an antidepressant medication or major tranquilizer at therapeutic doses for depression or psychosis for at least 3 months, a suicidal attempt, hospitalization for psychiatric disease, or a period of disability due to a psychiatric disease.
* History of immunologically mediated disease (e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hemolytic anemia, scleroderma, severe psoriasis, rheumatoid arthritis).
* History or other evidence of chronic pulmonary disease associated with functional limitation. Severe cardiac disease (e.g., NYHA Functional Class III or IV, myocardial infarction within 6 months, ventricular tachyarrhythmias requiring ongoing treatment, unstable angina or other significant cardiovascular diseases).
* History of a severe seizure disorder or current anticonvulsant use.
* Evidence of an active or suspected cancer or a history of malignancy where the risk of recurrence is >=20% within 2 years. Patients with a lesion suspicious of hepatic malignancy on a screening imaging study will only be eligible if the likelihood of carcinoma is <=10% following an appropriate evaluation.
* History of having received any systemic anti-neoplastic (including radiation) or immunomodulatory treatment (including systemic corticosteroids) <=6 months prior to the first dose of study drug or the expectation that such treatment will be needed at any time during the study.
* Major organ transplantation.
* Thyroid disease with thyroid function poorly controlled on prescribed medications. Patients with abnormal thyroid stimulating hormone or T4 concentrations, with elevation of antibodies to thyroid peroxidase and any clinical manifestations of thyroid disease are excluded.
* History or other evidence of severe retinopathy (e.g. CMV retinitis, macula degeneration) or clinically relevant ophthalmological disorder due to diabetes mellitus or hypertension
* Inability or unwillingness to provide informed consent or abide by the requirements of the study.
* History or other evidence of severe illness or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study.
* Patients with a value of alpha-fetoprotein >100 ng/mL are excluded, unless stability (less than 10% increase) has been documented over at least the previous 3 months.
* Evidence of drug and/or alcohol abuse (20g/day for women & 30g/day for men).
* Patients included in another trial or having been given investigational drugs within 12 weeks prior to screening
* Any known history of hypersensitivity to interferon.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-06; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Sustained response (HBeAg seroconversion and HBV DNA <2000 IU/ml) | 24 weeks post-treatment

SECONDARY OUTCOMES:
HBeAg loss and seroconversion | 24 weeks post-treatment and follow up for 5 years.
HBsAg loss and seroconversion | 24 weeks post-treatment and follow up for 5 years.
HBV DNA <2000IU/ml and undetectable | 24 weeks post-treatment and follow up for 5 years.
ALT normalization | 24 weeks post-treatment and long-term follow-up
Sustained response | 5 years post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Henry LY Chan, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

REFERENCES:
- [Background] Sung JJ, Tsoi KK, Wong VW, Li KC, Chan HL. Meta-analysis: Treatment of hepatitis B infection reduces risk of hepatocellular carcinoma. Aliment Pharmacol Ther. 2008 Nov 1;28(9):1067-77. doi: 10.1111/j.1365-2036.2008.03816.x. Epub 2008 Jul 24. PMID 18657133
- [Background] European Association For The Study Of The Liver. EASL clinical practice guidelines: Management of chronic hepatitis B virus infection. J Hepatol. 2012 Jul;57(1):167-85. doi: 10.1016/j.jhep.2012.02.010. Epub 2012 Mar 20. No abstract available. PMID 22436845
- [Background] Fung J, Lai CL, Tanaka Y, Mizokami M, Yuen J, Wong DK, Yuen MF. The duration of lamivudine therapy for chronic hepatitis B: cessation vs. continuation of treatment after HBeAg seroconversion. Am J Gastroenterol. 2009 Aug;104(8):1940-6; quiz 1947. doi: 10.1038/ajg.2009.200. Epub 2009 May 19. PMID 19455108
- [Background] Liang Y, Jiang J, Su M, Liu Z, Guo W, Huang X, Xie R, Ge S, Hu J, Jiang Z, Zhu M, Wong VW, Chan HL. Predictors of relapse in chronic hepatitis B after discontinuation of anti-viral therapy. Aliment Pharmacol Ther. 2011 Aug;34(3):344-52. doi: 10.1111/j.1365-2036.2011.04738.x. Epub 2011 Jun 14. PMID 21671967
- [Background] Wong VW, Wong GL, Yan KK, Chim AM, Chan HY, Tse CH, Choi PC, Chan AW, Sung JJ, Chan HL. Durability of peginterferon alfa-2b treatment at 5 years in patients with hepatitis B e antigen-positive chronic hepatitis B. Hepatology. 2010 Jun;51(6):1945-53. doi: 10.1002/hep.23568. PMID 20209602
- [Background] Marcellin P, Bonino F, Lau GK, Farci P, Yurdaydin C, Piratvisuth T, Jin R, Gurel S, Lu ZM, Wu J, Popescu M, Hadziyannis S; Peginterferon alfa-2a in HBeAg-negative Chronic Hepatitis B Study Group. Sustained response of hepatitis B e antigen-negative patients 3 years after treatment with peginterferon alpha-2a. Gastroenterology. 2009 Jun;136(7):2169-2179.e1-4. doi: 10.1053/j.gastro.2009.03.006. Epub 2009 Mar 19. PMID 19303414
- [Background] Song BC, Suh DJ, Lee HC, Chung YH, Lee YS. Hepatitis B e antigen seroconversion after lamivudine therapy is not durable in patients with chronic hepatitis B in Korea. Hepatology. 2000 Oct;32(4 Pt 1):803-6. doi: 10.1053/jhep.2000.16665. PMID 11003626
- [Background] Dienstag JL, Cianciara J, Karayalcin S, Kowdley KV, Willems B, Plisek S, Woessner M, Gardner S, Schiff E. Durability of serologic response after lamivudine treatment of chronic hepatitis B. Hepatology. 2003 Apr;37(4):748-55. doi: 10.1053/jhep.2003.50117. PMID 12668966
- [Background] Ryu SH, Chung YH, Choi MH, Kim JA, Shin JW, Jang MK, Park NH, Lee HC, Lee YS, Suh DJ. Long-term additional lamivudine therapy enhances durability of lamivudine-induced HBeAg loss: a prospective study. J Hepatol. 2003 Oct;39(4):614-9. doi: 10.1016/s0168-8278(03)00394-5. PMID 12971973
- [Background] van Nunen AB, Hansen BE, Suh DJ, Lohr HF, Chemello L, Fontaine H, Heathcote J, Song BC, Janssen HL, de Man RA, Schalm SW. Durability of HBeAg seroconversion following antiviral therapy for chronic hepatitis B: relation to type of therapy and pretreatment serum hepatitis B virus DNA and alanine aminotransferase. Gut. 2003 Mar;52(3):420-4. doi: 10.1136/gut.52.3.420. PMID 12584227